CLINICAL TRIAL: NCT04086056
Title: A Monocentric, Prospective Clinical Study to Evaluation of Cerebral Oxygen Saturation by Near InfraRed Spectroscopy (NIRS) in Children With Craniosynostosis
Brief Title: CraNIRS Clinical Study
Acronym: CraNIRS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0568; 2019-A02390-57 (Other: ID-RCB)
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Craniosynostoses
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with craniosynostosis: Children with craniosynostosis who will be operated in prone position.
  Interventions: Other: NIRS monitoring

INTERVENTIONS:
Other: NIRS monitoring — Regional cerebral oxygen saturation (rScO₂) will be collected by NIRS monitoring before anesthesia induction, during surgery and after extubation, in children with craniosynostosis.

SUMMARY:
Craniosynostosis is a rare disorder characterized by a premature fusion of one or more sutures of the skull. Craniosynostosis is usually diagnosed in the first years of life. Several complications may be identified if untreated, notably, developmental delay, and vision problems.

In some patients with craniosynostosis a decrease in cerebral blood perfusion can be identified. It might be related to the constriction of the brain caused by premature sutural fusion or the localized constriction of venous sinuses.

In this study the investigator use the NIRS which is defined as a non-invasive technique to monitor hemodynamic parameters and hemoglobin oxygen saturation of the brain during the surgical correction of the craniosynostosis. By applying this method the investigator will be able to analyse the changes in cerebral hemoglobin oxygen saturation related to the modification of the skull.

Determining changes in brain oxygen saturation by using NIRS before, during and after surgery will help both to better understanding the impact of surgical decompression on improving cerebral oxygenation and to better adapt anaesthesia strategies during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls.
* Aged 3 to 18 months old.
* Subjects with a craniosynostosis diagnosis confirmed by imaging.
* Craniosynostosis requiring a corrective surgery in ventral position.
* Parents/ legal guardian must provide non opposition prior to participation in the study.

Exclusion Criteria:

- Craniosynostosis planned to be corrected by an endoscopic craniectomy or in dorsal position.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with craniosynostosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Regional cerebral oxygen saturation measure | Day 0 before anesthesia
  Variations of rScO₂ (%, frequency of desaturations) measured by NIRS captors
Regional cerebral oxygen saturation measure | Day 0 during surgery
  Variations of rScO₂ (%, frequency of desaturations) measured by NIRS captors
Regional cerebral oxygen saturation measure | Day 0 after extubation
  Variations of rScO₂ (%, frequency of desaturations) measured by NIRS captors

CONTACTS AND LOCATIONS:
Overall Officials: Federico DI ROCCO, Principal Investigator — Hospices Civils de Lyon service neurochirurgie pédiatrique
Locations (1):
- Hospices Civils de Lyon service neurochirurgie pédiatrique, Bron, France